CLINICAL TRIAL: NCT06302296
Title: Evaluating the Effect of Injectable Platelet-rich Fibrin on Accelerating Orthodontic Tooth Movement During Leveling and Alignment Stage Study Description
Brief Title: Evaluating the Effect of Injectable Platelet-rich Fibrin on Accelerating Orthodontic Tooth Movement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hama University (Other)
Responsible Party: Principal Investigator, FADI JNAID, Syria-Hama University, Hama University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hama University/
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Tooth Mobility; Injectable Platelet-rich Fibrin
MeSH Terms: conditions — Tooth Mobility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- injectable form of PRF (Experimental): A group of patients in which participants will be undergo to orthodontic treatment will be received a 0.9 ml injection of PRF after 1st premolar extraction.
  Interventions: Device: injectable form of PRF
- traditional orthodontic treatment (Experimental): A group of patients in which participants will be undergo to traditional orthodontic treatment will be received a Placebo injection after 1st premolar extraction.
  Interventions: Behavioral: Placebo injection

INTERVENTIONS:
Device: injectable form of PRF — A group of patients in which participants will be undergo to orthodontic treatment will be received a 0.9 ml injection of PRF after 1st premolar extraction.
  Arms: injectable form of PRF
Behavioral: Placebo injection — A group of patients in which participants will be undergo to traditional orthodontic treatment will be received a Placebo injection after 1st premolar extraction.
  Arms: traditional orthodontic treatment

SUMMARY:
One of the main goals of orthodontic treatment is the reduction of treatment time through faster tooth movement. The previous studies evaluating platelet-rich fibrin (PRF) and orthodontic tooth movement (OTM) are limited, which makes the results difficult to generalize.

DETAILED DESCRIPTION:
One of the main goals of orthodontic treatment is the reduction of treatment time through faster tooth movement. The previous studies evaluating platelet-rich fibrin (PRF) and orthodontic tooth movement (OTM) are limited, which makes the results difficult to generalize. To this end, we set up this Randomized experiment to evaluate the effect of the injectable form of PRF (i-PRF) on OTM, using nonadditive containing i-PRF, which has higher levels of regenerative cells and growth factors compared with other PRF types because of the use of low centrifugation spee. Accordingly, we aimed to evaluate the effect of i-PRF on the rate of maxillary incisors leveling during comprehensive orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age (18-26). Severe or very severe irregularity of the upper incisors greater than (7 mm) according to Little's index, so it is recommended to extract the upper first premolar.

  * Class I or Class II malocclusion, first model according to Angle, with skeletal class I or II and a normal or mild vertical growth pattern.
  * All permanent upper teeth, up to the first molar, are present, with the possibility of attaching brackets to all teeth in a correct position.
  * The patient has good oral health.

Exclusion Criteria:

* • The presence of any systemic disease that affects orthodontic dental movement.

  * Severe malalignment of one of the teeth (palatal quadrant, ectopic canine, ectopic premolar).
  * The patient has undergone previous orthodontic treatment.
  * The patient is subject to any drug treatment that may affect orthodontic dental movement (cortisone, non-steroidal anti-inflammatory drugs).
  * The patient has poor oral health.
  * Commitment to periodic follow-up appointments.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Leveling and alignment maxillary incisors | One month ,two month,six month
  - Alginate impressions were taken at insertion of the first archwire (0.014-in nickel-titanium) maxillary incisors Leveling and alignment.
  Leveling and alignment were achieved through the following sequence of archwires: 0.014-in nickel-titanium (NiTi), 0.016 × 0.022-in NiTi, 0.017 × 0.025-in NiTi, 0.019 × 0.025-in stainless steel (SS)(3).

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Salami, MSc student, Principal Investigator — Hama University; Rabab Alsabbagh, Professor, Study Chair — Hama University
Locations (1):
- Fadi Jnaid, Hama, Syria

IPD SHARING:
Plan to Share IPD: No